CLINICAL TRIAL: NCT04981106
Title: The Effects of Elastic Band Exercise on the Pain, Kinesiophobia, Functional, and Psychological Status After Total Knee Arthroplasty
Brief Title: Elastic Band Exercise on the Pain, Kinesiophobia, Functional, and Psychological Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Funda Cetinkaya, Associate Professor Doctor, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/08-16
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Exercise
Keywords: elastic band exercise; kinesiophobia; functional, psychological status
MeSH Terms: conditions — Motor Activity; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Band Exercise (Experimental): All the participants were subjected to walking training and a standard postoperative care and exercise protocol until discharged from the hospital. During discharging, all the participants in both groups were provided with explanation and illustration about how to perform the exercises. In order to prevent any problem, the participants in both groups were recommended to start the at-home rehabilitation programs, which incorporate knee movement exercises, to be ready 2 weeks (14 days) after the surgery and they were asked to continue their current exercise programs thus far.
  The patients in intervention group were recommended to do, in addition to the at-home exercise program given to the patients in control group, elastic band exercises and researchers showed them how to use the elastic bands by making use of instructions.
  Interventions: Other: Elastic Band Exercise
- Exercise (No Intervention): The patients in control group were recommended to maintain only an at-home exercise program incorporating knee flexion and extension exercises.

INTERVENTIONS:
Other: Elastic Band Exercise — The participants were asked to do exercise 4 times a day with a minimum of 2 hours interval between the sessions. The participants were instructed to avoid elastic band exercise 1 hour before or after the meals in order to prevent a physical impairment and to adopt a moderately progressive approach in order to prevent lower extremity pain after exercise and to increase the sense of success and confidence.
  Through phone calls, researchers asked the participants in intervention group if they do the elastic band exercises at home and if they had any difficulty while doing these exercises, as well as the reasons if they haven't done the exercises. When the participants in control and intervention groups returned to hospital after 4 weeks, the knee joint movement, lower extremity strength, knee joint pain, quality of life, kinesiophobia, and depression levels and physical functions of these groups were compared.
  Arms: Elastic Band Exercise

SUMMARY:
Aiming to determine the effects of elastic band exercise on kinesiophobia, functional capacity, and depression after the total knee arthroplasty, the present study was designed and carried out as a randomized controlled trial study. The study was carried out between October 2019 and April 2020 in the Physical Therapy and Rehabilitation Department of a training and research hospital.This study, the effects of elastic band exercise program on the pain, kinesiophobia, quality of life, depression, and functional capacity of TKA patients were examined. Elastic band exercise program significantly decreased the pain level, exercise fear, and depression level of patients and positively contributed to the quality of life and functional capacity.

DETAILED DESCRIPTION:
All the participants were subjected to walking training and a standard postoperative care and exercise protocol until discharged from the hospital. During discharging, all the participants in both groups were provided with explanation and illustration about how to perform the exercises. In order to prevent any problem, the participants in both groups were recommended to start the at-home rehabilitation programs, which incorporate knee movement exercises, to be ready 2 weeks (14 days) after the surgery and they were asked to continue their current exercise programs thus far. The patients in control group were recommended to maintain only an at-home exercise program incorporating knee flexion and extension exercises.

The patients in intervention group were recommended to do, in addition to the at-home exercise program given to the patients in control group, elastic band exercises and researchers showed them how to use the elastic bands by making use of instructions.The participants were asked to do exercise 4 times a day with a minimum of 2 hours interval between the sessions. The participants were instructed to avoid elastic band exercise 1 hour before or after the meals in order to prevent a physical impairment and to adopt a moderately progressive approach in order to prevent lower extremity pain after exercise and to increase the sense of success and confidence.

ELIGIBILITY:
Inclusion Criteria:

Unilateral Total Knee Arthroplasty

Exclusion Criteria:

Bilateral Total Knee Arthroplasty

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Tampa kinesiophobia index | First measurement two weeks after surgery (intervetion 58.2; control 54.1)
  Tampa is a 17-item scale
WOMAC Osteoarthritis Index | First measurement two weeks after surgery (intervetion 89.3; control 88.1)
  WOMAC is a valid and reliable index that is widely used for assessing the patients with osteoarthritis.
Beck's Depression Inventory | First measurement two weeks after surgery (intervetion 21.6; control 22.1)
  21 items in total.

SECONDARY OUTCOMES:
Tampa kinesiophobia index | Second measurement six weeks after surgery (intervetion 36.9; control 42.9)
  Tampa is a 17-item scale
WOMAC Osteoarthritis Index | Second measurement six weeks after surgery (intervetion 29; control 70.5)
  WOMAC is a valid and reliable index that is widely used for assessing the patients with
Beck's Depression Inventory | Second measurement six weeks after surgery (intervetion 6.9; control 13.2)
  21 items in total.

CONTACTS AND LOCATIONS:
Overall Officials: Funda CETINKAYA, Principal Investigator — Aksaray University; Ahmet KARAKOYUN, Dr, Principal Investigator — Aksaray University
Locations (1):
- Funda CETINKAYA, Aksaray, Select State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cetinkaya F, Karakoyun A. The effects of elastic band exercise on the pain, kinesiophobia, functional, and psychological status after total knee arthroplasty: a randomized controlled trial. Clin Rheumatol. 2022 Oct;41(10):3179-3188. doi: 10.1007/s10067-022-06266-0. Epub 2022 Jul 1. PMID 35776283